CLINICAL TRIAL: NCT00006474
Title: Phase I Trial of Temodar Plus O6-Benzylguanine (O6-BG) (NSC 637037) in the Treatment of Patients With Newly Diagnosed (Part 1) or Recurrent/Progressive (Parts 1 and 2) Cerebral Anaplastic Gliomas
Brief Title: Temozolomide and O6-benzylguanine in Treating Patients With Newly Diagnosed, Recurrent, or Progressive Anaplastic Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1388; DUMC-1388-02-8R2; DUMC-1388-00-8; NCI-490; DUMC-1388-01-8R1; CDR0000068301 (Other: DUMC)
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — O(6)-benzylguanine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: temozolomide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining temozolomide and O6-benzylguanine in treating patients who have newly diagnosed, recurrent, or progressive anaplastic glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of O6-benzylguanine (O6-BG) effective in producing complete suppression of tumor O6-alkylguanine-DNA alkyltransferase activity in patients with newly diagnosed (closed to accrual 12/19/2000) or recurrent or progressive cerebral anaplastic glioma.
* Determine the maximum tolerated dose of temozolomide administered after O6-BG in these patients.
* Determine the toxicity of this regimen in these patients.
* Determine the anti-tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

* Part I: Patients receive escalating doses of O6-benzylguanine (O6-BG) IV continuously for 49 hours until the dose that produces the target depletion of tumor O6-alkylguanine-DNA alkyltransferase (AGT) is determined. Patients undergo a craniotomy after completion of the O6-BG infusion. (closed to accrual 12/19/2000)
* Part II: After determination of the O6-BG dose in Part I, patients with recurrent malignant gliomas receive O6-BG IV continuously for 49 hours beginning on day 1. Patients also receive oral temozolomide on day 1. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 20-30 patients (with 14 patients participating in Part II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Part I:

  * Histologically confirmed, newly diagnosed glioblastoma multiforme or anaplastic astrocytoma (closed to accrual 12/19/2000)
* Parts I and II:

  * Histologically confirmed astrocytic, oligodendroglial, or mixed glial tumor

    * Grade III or higher
    * Recurrent or progressive after radiotherapy
* Evaluable residual disease by contrast-enhanced MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* SGOT no greater than 2.5 times upper limit of normal
* Bilirubin normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* BUN no greater than 25 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 weeks since prior biologic therapy and recovered

Chemotherapy:

* At least 2 weeks since prior chemotherapy (including but not limited to topotecan) and recovered

  * Patients in trials with one of the following treatment combinations are allowed to enroll 6 weeks after receiving carmustine (BCNU):

    * BCNU on day 1
    * BCNU on day 1 and topotecan on days 1, 8, 15, 22, 29, and 36
    * BCNU on day 1 and irinotecan on days 1, 8, 15, and 22

Endocrine therapy:

* Patients on corticosteroids must be on a stable dose for at least 2 weeks before study
* At least 6 weeks since other prior endocrine therapy and recovered

Radiotherapy:

* See Disease Characteristics
* At least 6 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Quinn JA, Jiang SX, Reardon DA, Desjardins A, Vredenburgh JJ, Rich JN, Gururangan S, Friedman AH, Bigner DD, Sampson JH, McLendon RE, Herndon JE Jr, Walker A, Friedman HS. Phase I trial of temozolomide plus O6-benzylguanine 5-day regimen with recurrent malignant glioma. Neuro Oncol. 2009 Oct;11(5):556-61. doi: 10.1215/15228517-2009-007. Epub 2009 Mar 16. PMID 19289491
- [Result] Quinn JA, Desjardins A, Weingart J, Brem H, Dolan ME, Delaney SM, Vredenburgh J, Rich J, Friedman AH, Reardon DA, Sampson JH, Pegg AE, Moschel RC, Birch R, McLendon RE, Provenzale JM, Gururangan S, Dancey JE, Maxwell J, Tourt-Uhlig S, Herndon JE 2nd, Bigner DD, Friedman HS. Phase I trial of temozolomide plus O6-benzylguanine for patients with recurrent or progressive malignant glioma. J Clin Oncol. 2005 Oct 1;23(28):7178-87. doi: 10.1200/JCO.2005.06.502. PMID 16192602